CLINICAL TRIAL: NCT06868407
Title: Randomized Control Trial of Electronic, Self-Guided Safety Plan in Adolescents: Project SAFER
Brief Title: Electronic, Self-Guided Safety Plan in Adolescents: Project SAFER
Acronym: Project SAFER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Responsible Party: Principal Investigator, Kathryn Fox, Assistant Professor, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2200661-2; 2200661-2 (Other: DU IRBnet number)
Record Dates: First submitted 2025-02-19; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Suicide Attempt; Suicide Ideation
Keywords: adolescent; suicide; safety plan intervention; RCT
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 fashion to either the electronic, self-guided safety plan or the psychoeducational control.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Random assignment to condition will be conducted in a triple-masked manner. Participants will be masked to whether they received active treatment and investigators will be masked to which condition the participant is randomized to-as the randomization occurs automatically within the Qualtrics survey. Additionally, as the primary and secondary outcomes are self-report measures, we will not be utilizing an outcomes assessor (e.g. a clinical interviewer).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Guided Electronic Safety Plan Intervention (Experimental): Participants in this arm are assigned to the electronic, self-guided safety plan.
  Interventions: Behavioral: Experimental: Self-Guided Electronic Safety Plan Intervention
- Psychoeducation about Suicide Crisis Resources (Control Intervention) (Active Comparator): Participants in this arm are assigned to the active control intervention

INTERVENTIONS:
Behavioral: Psychoeducation about Suicide Crisis Resources (Control Intervention) — The active control intervention includes psychoeducation about suicide crisis services, with a particular focus on breaking down myths and barriers to using suicide crisis services use.
Behavioral: Experimental: Self-Guided Electronic Safety Plan Intervention — This is a modified version of the E-SPI first created by Methi and colleagues (2024) which was originally adapted from the six primary steps of the Stanely-Brown safety plan (identifying warning signs, internal coping strategies, social distractions, non-professional crisis contacts, professional crisis resources, suicidal means restriction). Modifications to the E-SPI were based on pilot-study participant feedback and feedback from a youth focus group. The intervention was updated in accordance with pilot-study participant feedback and feedback from subsequent youth interviews. Modification examples include updated instruction wording to reduce ambiguity, updated illustrations, and increased accessibility for participants with reading-based learning disabilities.
  Other Names: E-SPI
  Arms: Self-Guided Electronic Safety Plan Intervention

SUMMARY:
Suicide is a leading cause of death for youth 10-24, and nearly ¼ of adolescents report nonfatal suicidal thoughts and behaviors (STB). However, traditional interventions (e.g., multi-session therapy protocols) are contingent upon (1) access to treatment, (2) involvement of parents/guardians (hereafter parents), and (3) disclosure of risk to treatment providers. Unfortunately, adolescents are frequently hesitant to disclose STB to healthcare providers and parents for reasons including shame, stigma, and fear of hospitalization, with even lower rates of disclosure among queer youth-including those with diverse genders and sexualities- who are at disproportionately high risk for STB. Related to these concerns, most youth at risk for suicide, as well as other mental health challenges, do not access any mental healthcare. Self-guided, brief digital interventions may be a powerful adolescent suicide prevention tool. With their relative accessibility-they can be completed privately, at home, for at no cost-such interventions are well-suited for youth not accessing traditional care. Thus, effective digital adaptation of brief suicide prevention interventions is a promising frontier for adolescent suicide prevention.

A strong candidate for digital adaptation is the Safety Planning Intervention (SPI), a brief (~5-10 minute) single-session intervention shown to significantly reduce STB in adults. In the SPI, people at risk for suicide receive brief education about suicidal thoughts and crises before developing a personalized, one-page plan with skills and resources to use during future suicide crises, when it is difficult to think clearly. There is strong evidence across several randomized control trials (RCTs) that SPI reduce suicidal behaviors in adults compared to those who received treatment as usual. Despite widespread use in outpatient and acute clinical settings across ages, there is a paucity of adequately-powered RCTs testing whether the SPI (in any format) reduces STB in adolescents.

Emerging evidence supports the SPI can work well in digital format among adolescents. In qualitative studies, adolescents with a history of STBs reported that they would be comfortable using a digital safety plan and feel it would be helpful to them in a crisis, emphasizing easy access and customizability as useful features. Building on this work, I created a digital, self-guided SPI specifically for use in online studies of high-risk adolescents. Preliminary research (approved by DU IRB# 1505797) suggests that youth find this self-guided digital SPI "very helpful" and nearly half actually use the safety plan in the next month. Moreover, using a standardized coding system, quality of self-guided safety plans mirrored the quality seen in clinician-guided, adult SPI. However, it remains unclear whether the SPI in any format can reduce STB in adolescents.

This project will test the ability of a self-guided SPI, compared to a suicide psychoeducational control intervention, to increase self-efficacy to avoid suicidal behaviors and to reduce suicidal thoughts and suicidal behaviors in adolescents over a 3-month follow-up period. The investigators hypothesize that compared to the control condition, adolescents who receive the SPI will report greater self-efficacy to avoid suicidal action and reduced STB at the 3-month follow-up assessment. If hypotheses are supported, this study will provide strong, high-quality evidence in favor of the potential of highly accessible, digital self-guided SPIs to prevent suicidal behavior in adolescents. In this case, distribution of such an intervention at scale could be a powerful tool for reducing STBs in adolescents.

DETAILED DESCRIPTION:
Participants will be recruited via advertisements posted primarily online to web-based forums and social media (e.g., discord, Instagram). Digital recruitment flyers will also be distributed to youth-serving organizations and mental health clinics to share with the adolescents they serve. In communications with participants, the investigators will call this study "Project SAFER." Those who see study ads and are interested in participating will be directed to click the hyperlink directing them to Qualtrics where they will complete an eligibility survey assessing inclusion/exclusion criteria for the study (see attached).

Individuals who qualify will be shown a study assent form delineating all study components. Those who "agree" to participate will then complete a brief quiz to ensure they understand the risks and benefits of participating. Individuals who do not qualify for the studies will be notified that they do not qualify, and they will be provided with electronic mental health resources. Participants will be told they can take the quiz up to 3 times before they will be told they do not qualify.

All aspects of the study be completed online, via Qualtrics.

There are two primary parts of the study:

1. Part 1 (~30 minutes): Participants will complete the baseline survey, before being randomized to either the electronic self-guided intervention or psychoeducational control intervention. Finally, participant will post intervention measures.
2. Part 2 (~15 minutes): Three months after part 1, participants will be contacted to complete Part 2, assessing suicidal thoughts and behaviors and other key outcomes, since completing Part 1.

Halfway through the follow-up period (1.5 months after completing Part 1), participants will receive a follow-up message reminding them about their safety plan (treatment group) or resource list (control group). Finally, all participants in the control group will be offered the Safety Plan at the end of Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English
* Internet access,
* Past-month suicidal thoughts AND a past-year suicide attempt OR at least 5 days of suicidal thoughts in the past year.

Exclusion Criteria:

* disability that interferes with the ability to complete the study on a computer
* not in US
* response that indicates bot or fraudulent

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Average scores on self-efficacy to avoid future suicidal action score | Post-intervention AND across 3-month follow-up period
  Responses to a question measuring self-efficacy to avoid future suicidal behavior: "If you have serious thoughts of killing yourself in the future, how confident are you that you WILL BE ABLE to keep yourself from attempting suicide?" (Czyz et al., 2016)
Average perceived suicide-related coping capacity | immediately post intervention AND across 3-month follow-up period
  Average scores on a composite of 3 items from the Stanley et al. 2017 measure of suicide-related coping (i.e., I have several things I can do to get through a suicidal crisis, I do not think there is anything that I can do to help myself when I am feeling suicidal (R), I am at the mercy of my suicidal thoughts (R))

SECONDARY OUTCOMES:
Days of suicide ideation over 3 month period | 3 months
  Self-reported days of suicide ideation over the 3 month follow-up period using the SITBI-R (Fox et al., 2020)
Number of participants reporting suicidal behaviors over follow-up | 3 months
  Number of participants reporting engagement (presence/absence) in suicidal behaviors (suicide attempt, aborted attempt, interrupted attempt) over the 3 month follow-up period using the SITBI-R (Fox et al., 2020)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Fox, PhD, Principal Investigator — University of Dener
Locations (1):
- University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be collected online (single site), via Qualtrics, an encrypted and HIPAA-compliant platform. Our Qualtrics Surveys will be shared across study team members at University of Denver. Recruitment and participation will be monitored by members of the study team.
  When the study is completed: Data will downloaded from Qualtrics and will be stored on HIPAA compliant servers (smb://shares.du.edu/research/AHSS Psychology/Fox Lab) rather than individual computers. De-identified data (data WITHOUT email addresses, phone numbers, etc) will be kept indefinitely and may be made available to other researchers for other studies following the completion of this research study (e.g., on osf.io). For example, when the research is completed, anonymized data may be saved for use in future research and may be posted online (e.g., posted on osf.io).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 1 year after completing data collection OR upon submission of the manuscript to a peer-reviewed journal. The data will be available open access thereafter.
Access Criteria: The de-identified data will be shared open access